CLINICAL TRIAL: NCT04254562
Title: Helping Youth on the Path to Employment: Creating Economic Self-sufficiency
Brief Title: Helping Youth on the Path to Employment
Acronym: HYPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Colorado State University (Other); National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency); Binghamton University (Other)
Responsible Party: Principal Investigator, Michelle Mullen, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H00017845; HHS-2019-ACL-NIDILRR-RTEM-0334 (Other Grant/Funding Number: NIDILRR)
Record Dates: First submitted 2020-01-15; First posted 2020-02-05 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-03

CONDITIONS: Mental Impairment; Educational Problems
Keywords: Supported Employment; Supported Education; Mental Health; Behavioral Health; Cognitive Remediation
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group: HYPE Services (Experimental): The experimental arm will receive the HYPE intervention for 12 months.
  Interventions: Behavioral: Weekly Meetings with a Supported Employment/Supported Education Specialist; Behavioral: Focused Skill and Strategy Training (FSST)
- Control Group: Enhanced Academic Services as Usual (Active Comparator): The control arm will receive a special personalized packet of resources available on campus and off-campus within a 10-mile radius, as "enhanced academic services as usual."
  Interventions: Behavioral: Enhanced Services as Usual

INTERVENTIONS:
Behavioral: Weekly Meetings with a Supported Employment/Supported Education Specialist — Participants will receive intervention for 12 months which includes weekly meetings with a Supported Employment/Supported Education Specialist (HYPE Specialist). During the weekly meetings, the HYPE Specialist will review each participant's education and employment goals, and deliver individualized support relevant to those goals which include use of structured HYPE tools and worksheets as needed.
  Arms: Experimental Group: HYPE Services
Behavioral: Focused Skill and Strategy Training (FSST) — Participants receive a 12 week Focused Skill and Strategy Training (FSST), a structured cognitive remediation intervention.
  Arms: Experimental Group: HYPE Services
Behavioral: Enhanced Services as Usual — One hour meetings every semester to review individual academic needs and review list of available on campus resources to best meet the student's needs.
  Arms: Control Group: Enhanced Academic Services as Usual

SUMMARY:
Helping Youth on the Path to Employment (HYPE): Creating economic self-sufficiency, a randomized-controlled implementation efficacy hybrid trial, will test a manualized intervention combining educational and employment supports for young adults with mental health conditions on a college campus.

DETAILED DESCRIPTION:
Previous controlled trials in mature adult subjects has consistently demonstrated that Supported Employment interventions (i.e., Individual Placement and Supports) elicit benefit for those with mental health conditions in getting and keeping productive work. Similarly, previous research demonstrates that Supported Education has efficacy in helping young adults with mental health conditions in their academics. However, to date, no evidence-based practice exists which combines both supported education and supported employment interventions into a single model that has efficacy and utility for young adults with serious mental health conditions. Supported Education has been fruitful for navigating academics, but hasn't demonstrated efficacy for supporting young adults with their careers, and Supported Employment programs, like IPS, have shown poor efficacy for helping young adults, as it was designed to assist mature adults. Therefore, the HYPE Model will become the first evidence-informed intervention to combine Supported Employment and Supported Education paradigms in an effort to help young adults with mental health conditions successfully navigate college so they can move into a primary labor market career and attain economic self-sufficiency. Furthermore, this study will be employed from within the university setting itself, on the college campus, and will be embedded directly in either Services for Students with Disabilities (SSD) (i.e., Office of disability services) or Office of Counseling Services.

ELIGIBILITY:
Inclusion Criteria:

* be between 18-30 years of age
* able to speak and read English fluently
* cognitively capable of providing informed consent and participating in study activities;
* enrolled in a minimum of six credits at a campus-based accredited college (two year or four-year programs)
* intending to enroll in a minimum of four semesters of college courses with the expectation of being continuously enrolled
* have had at least one prior academic disruption during a college academic semester - (e.g., withdrawal from postsecondary institutions; academic probation; not meeting satisfactory academic progress; or a prior leave of absence) prior to study enrollment
* currently have a diagnosed mental health condition by a licensed mental health provider under the DSM-V Axis 1 diagnoses (schizophrenia or other psychotic disorders, anxiety disorders, mood disorders, eating disorders, attention deficits and disruptive behavior disorders) or have been deemed eligible for ADA protections due to a disabling mental health condition - (e.g., receiving state vocational agency services, SSI/DI benefits, or postsecondary accommodations).

Exclusion Criteria:

* have received or are receiving supports consistent with HYPE in the past year;
* have had no impact to academic success in college (i.e. disruption);
* have a secondary autism spectrum disorder, traumatic brain injury, or other neurodevelopmental or neurocognitive disorder affecting cognition;
* are currently incarcerated prisoners;
* are unable to speak or read English fluently;
* are under age 18 or require a legal guardian to provide informed consent;
* lack the cognitive capability to provide informed consent on their own

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Number of students making satisfactory academic progress | 24 months
  Number of students making satisfactory academic progress (SAP), defined as a student completing two-thirds of the courses they enroll in each semester and achieving a GPA of 2.0 or greater
Number of students with disruptions toward completion of college degree. | 24 months
  Number of students with disruptions toward completion of college degree, defined as withdrawal from postsecondary institutions, academic probation, not meeting satisfactory academic progress, or a leave of absence

SECONDARY OUTCOMES:
Change in frequency of educational barriers | 24 months
  The average frequency of educational barriers experienced by participants, defined as the specific challenges participants face in their pursuit of postsecondary education and whether and how their use of accommodations through campus disability services has or would be helpful for them. This will be measured with the Educational Barriers Questionnaire.
Change in levels of perceived Stress | 24 months
  Change in levels of perceived stress throughout the study in the experimental condition, measured by the perceived stress scale.
Academic Self-Efficacy | 24 months
  Changes in academic self-efficacy among students across the study will be measured with the college self-efficacy scale and is defined as assess the degree to which participants' feel confident in their ability to complete tasks in college
Reliance on Social Security Benefits | 24 months
  Changes on students' reliance on Social Security benefits will be measured via self-report on the Baseline and Follow-up Demographics surveys

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Mullen, MS, Principal Investigator — UMass Medical School
Locations (3):
- United States (3):
  - Colorado State University, Fort Collins, Colorado
  - UMass Medical School, Worcester, Massachusetts
  - Binghamton University, Binghamton, New York

IPD SHARING:
Plan to Share IPD: Yes
Yes, individual deidentified participant data will be shared to ICPSR per funder (NIDILRR) regulations. Datasets will include: screening data (eligible participants only), baseline data, follow-up time 1 data, follow-up time 2 data, follow-up time 3 data, transcript data. Each dataset will share the same unique identifier (study ID) as well as date the data was collected. Codebooks (PDF format) and data dictionaries (CSV or TXT) will also be shared.
Supporting Information: Study Protocol
Time Frame: Data will be shared within 3 years of the completion of the study (estimated 2024-2027)
Access Criteria: If individuals outside of the study team (e.g. grad students) want data access they need to submit a formal request and if approved, be added to the IRB protocol & complete all necessary human subjects research certifications. They will be required to sign data use agreements. Any external researchers must sign a user agreement form before obtaining data. Data resulting from this project will be distributed at no cost. The user agreement is a UMMS requirement and this procedure is similar to those used by similar projects. The user agreement includes a detailed description of limitations on the redistribution/use of the data. External users are also required to limit publications to topics indicated in the agreement. Publications resulting from using data will reference the source as provided in agreement form; recommended citations will be provided. An investigator/Project Director will monitor dataset use to ensure data are handled properly and utilized for original purposes.